CLINICAL TRIAL: NCT01315509
Title: Dental Status of Patients With Severe Mental Illness
Acronym: SMI-DENTAL
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: DR. RENA COOPER-KAZAZ, HADASSAH MEDICAL ORGANIZATION
Other Study IDs: SMIDENTIST-HMO-CTIL
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Schizophrenia; Bipolar Disorder; PTSD; Depression
Keywords: Severe mental illness; Dental measures; Resistant depression
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Stress Disorders, Post-Traumatic; Depression; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The investigators aim to assess the dental status of psychiatric patients suffering from severe mental illness (schizophrenia, bipolar disorder, ptsd, resistant depression).

DETAILED DESCRIPTION:
PATIENTS WILL BE ASSESSED USING THE

1. DMFT (Decayed/Missing/Filled teeth)

AN EPIDEMILOGICAL ASSESSMENT TOOL THAT ASSESSES:

1. THE NUMBER OF TEETH WITH CURRENT DECAY
2. THE NUMBER OF TEETH MISSING
3. THE NUMBER OF TEATH TREATED IN THE PAST (FILLED)

2. CPI - Community Periodontal Index AN ASSESSMENT OF THE GUMS

3. OHIP-Oral Health Impact Profile A SELF-RATING FORM TO ASSESS THE SOCIAL AND FUNCTIONAL AFECTS OF THIER DENTAL STATUS

ELIGIBILITY:
Inclusion Criteria:

* All psychiatric patients suffering from schizophrenia, bipolar disorder, PTSD or resistant depression

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: THE SEVERE MENTAL ILL IN THE PSYCHIATRIC POPULATION OF THE HADASSAH MEDICAL ORGINIZATION -PSYCHIATRIC OUTPATIENT CLINIC
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2011-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rena Cooper-Kazaz, Israel, Israel

REFERENCES:
- [Background] Matevosyan NR. Oral health of adults with serious mental illnesses: a review. Community Ment Health J. 2010 Dec;46(6):553-62. doi: 10.1007/s10597-009-9280-x. Epub 2009 Dec 29. PMID 20039129